CLINICAL TRIAL: NCT04794179
Title: CROS and Quality of Life of Elderly Cochlear Implant Recipients and Their Care Givers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Advanced Bionics (Industry)
Responsible Party: Principal Investigator, Richard Gurgel, Principle Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00110953
Record Dates: First submitted 2019-02-01; First posted 2021-03-11 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Naida Link CROS device (Experimental): Individuals 18+ who already have Advanced Bionics CII/90K/Ultra cochlear implants will be given Naida Link CROS device to assess the effect the device has on speech understanding in challenging listening situations and on the quality of life in unilateral cochlear implant recipients and their frequent communication partners.
  Interventions: Device: Naida Link CROS

INTERVENTIONS:
Device: Naida Link CROS — Individuals 18+ who already have Advanced Bionics CII/90K/Ultra cochlear implants will be given Naida Link CROS device to assess the effect the device has on speech understanding in challenging listening situations and on the quality of life in unilateral cochlear implant recipients and their frequent communication partners.

SUMMARY:
The purpose of this study is to assess the effect of the Naida Link contralateral routing of signal (CROS) device on speech understanding in challenging listening situations and on the quality of life in unilateral CI recipients and their frequent communication partners. We hypothesize that:

1. Unilateral CI recipients will obtain higher speech understanding scores with the CROS device in challenging listening conditions
2. Use of the CROS device will lead to positive changes in ratings on Quality of Life measures for (i) unilateral CI recipients, and (ii) their frequent communication partners

A frequent communication partner (FCP) is an individual (a family member, or a friend, or a care taker, or a significant other, or a colleague, etc.) who has at least two hours of in-person interactions with the CI recipient every week.

DETAILED DESCRIPTION:
Cochlear Implants (CI) are now a well-accepted treatment for individuals with severe to profound hearing impairment. Compared to using one CI, bilateral CIs are known to provide access to some of the benefits of binaural hearing like improved speech understanding in noise (primarily due to headshadow), improved localization, reduced stress and fatigue, and improved quality of life (e.g., Dunn et al. 2012, Litovsky et al. 2012, Härkönen et al. 2016, Reeder et al. 2014, Agrawal 2008). However, a number of CI recipients are unable to or choose not to be implanted bilaterally for many reasons. Those with acoustic hearing in the contralateral ear can benefit significantly by using a hearing aid in that ear (bimodal hearing) (Ching et el. 2006, Dorman and Gifford 2010, Dorman et al. 2015, Dunn et al. 2005, Firszt et al. 2012, Illg et al. 2014, Farinetti et al. 2015).

Unilateral CI recipients do not have access to advantages of bilateral and bimodal hearing. In addition to reduced speech understanding in noise, especially when the speech source is located towards the non-CI, they can also experience increased stress and fatigue. Studies have shown that a CROS device, when worn on the contralateral, non-implanted ear, can help overcome speech understanding deficits due to head-shadow. The effect of such technology on quality of life of the CI recipient and their frequent communication partners has not been evaluated over an extended duration of use.

Study methodology:

Fourteen unilateral CI recipients will participate in this study. Testing will be conducted at the University of Utah Hospital ENT clinic. The study will comprise of 2 clinic visits separated by a take-home phase of 6 months. A designated FCP will be a part of each study visit, preferably.

Following are the test measures for CI recipients:

* Questionnaires
* Data logs
* Pure-tone audiometry
* Speech intelligibility

Following are the test measures for FCPs:

• Questionnaires

Speech testing will be conducted in a sound booth with a two speaker set-up (± 90°). AZBio sentences (Spahr et al., 2012) presented at 65 dB A will be the target stimuli. The interferer will be a multi-talker babble. The babble will be presented at an individualized level for each participant where their performance in noise in SCROS(Off)NCI configuration is half of their performance in quiet in SCROS(Off) configuration.

Study devices: For speech testing in the sound booth, a study Naida CI Q90 sound processor will be used. For the take-home phase, recipients will use their own Naida CI processor (Q70 or Q90). A Naida Link CROS will also be used for sound-booth testing as well as the take-home phase.

Workflow:

After recruiting, following will be mailed to the participants to be completed prior to the study visit and hand carried to visit 1:

For each CI subject:

(i) Informed consent form (ii) APS-SSD (Schafer et al, 2013, modified by H. Snapp, 2017) (iii) Nijmegen questionnaire (adapted from Hinderink et al, 2000)

For each CI subject's frequent communication partner:

(i) Informed consent form (ii) SOS-HEAR

ELIGIBILITY:
Inclusion Criteria:

* Unilateral recipients of Advanced Bionics CII/90K/Ultra implants
* Ages 18 years and above
* At least 6 months of CI use experience
* Current users of a Naida CI Q70 or Q90 processor
* Do not currently use a Naida Link CROS device
* Limited usable/aidable hearing in the contralateral ear
* Fluent in spoken English
* Willingness to use the CROS device regularly for the study duration
* Willingness to follow-up on a biweekly/monthly basis

Exclusion Criteria:

* < 6 months of CI use experience
* < 30% sentence recognition scores in quiet with unilateral CI
* Inability to participate in speech testing
* Inability to follow and complete questionnaires
* Inability to designate an FC
* not a unilateral recipient of Advanced Bionics CII/90K/Ultra implants

Frequent communication partner (FCP) participants' inclusion criteria:

* Ages 18 years and above
* Fluent in spoken English
* Willingness to participate in the study
* Spends at least two hours of in-person interactions with the recipient of Advanced Bionics CII/90K/Ultra implants every week.

FCP's Exclusion criteria:

* Under the age of 18 years
* Not fluent in spoken English
* Spends less than two hours of in-person interactions with the recipient of Advanced Bionics CII/90K/Ultra implants per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gurgel, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Heath, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal S. (2008) Spatial hearing abilities in adults with bilateral cochlear implants. PhD diss., University of Wisconsin-Madison.
- [Background] Ching TY, Incerti P, Hill M, van Wanrooy E. An overview of binaural advantages for children and adults who use binaural/bimodal hearing devices. Audiol Neurootol. 2006;11 Suppl 1:6-11. doi: 10.1159/000095607. Epub 2006 Oct 6. PMID 17063004
- [Background] Dorman MF, Cook S, Spahr A, Zhang T, Loiselle L, Schramm D, Whittingham J, Gifford R. Factors constraining the benefit to speech understanding of combining information from low-frequency hearing and a cochlear implant. Hear Res. 2015 Apr;322:107-11. doi: 10.1016/j.heares.2014.09.010. Epub 2014 Oct 5. PMID 25285624
- [Background] Dorman MF, Gifford RH. Combining acoustic and electric stimulation in the service of speech recognition. Int J Audiol. 2010 Dec;49(12):912-9. doi: 10.3109/14992027.2010.509113. Epub 2010 Sep 27. PMID 20874053
- [Background] Dunn CC, Tyler RS, Witt SA. Benefit of wearing a hearing aid on the unimplanted ear in adult users of a cochlear implant. J Speech Lang Hear Res. 2005 Jun;48(3):668-80. doi: 10.1044/1092-4388(2005/046). PMID 16197280
- [Background] Dunn CC, Tyler RS, Witt S, Ji H, Gantz BJ. Sequential bilateral cochlear implantation: speech perception and localization pre- and post-second cochlear implantation. Am J Audiol. 2012 Dec;21(2):181-9. doi: 10.1044/1059-0889(2012/12-0004). Epub 2012 Jul 30. PMID 22846635
- [Background] Farinetti A, Roman S, Mancini J, Baumstarck-Barrau K, Meller R, Lavieille JP, Triglia JM. Quality of life in bimodal hearing users (unilateral cochlear implants and contralateral hearing aids). Eur Arch Otorhinolaryngol. 2015 Nov;272(11):3209-15. doi: 10.1007/s00405-014-3377-8. Epub 2014 Nov 6. PMID 25373837
- [Background] Firszt JB, Holden LK, Reeder RM, Cowdrey L, King S. Cochlear implantation in adults with asymmetric hearing loss. Ear Hear. 2012 Jul-Aug;33(4):521-33. doi: 10.1097/AUD.0b013e31824b9dfc. PMID 22441359
- [Background] Harkonen K, Kivekas I, Rautiainen M, Kotti V, Sivonen V, Vasama JP. Sequential bilateral cochlear implantation improves working performance, quality of life, and quality of hearing. Acta Otolaryngol. 2015 May;135(5):440-6. doi: 10.3109/00016489.2014.990056. Epub 2015 Feb 13. PMID 25677966
- [Background] Illg A, Bojanowicz M, Lesinski-Schiedat A, Lenarz T, Buchner A. Evaluation of the bimodal benefit in a large cohort of cochlear implant subjects using a contralateral hearing aid. Otol Neurotol. 2014 Oct;35(9):e240-4. doi: 10.1097/MAO.0000000000000529. PMID 25058838
- [Background] Litovsky RY, Goupell MJ, Godar S, Grieco-Calub T, Jones GL, Garadat SN, Agrawal S, Kan A, Todd A, Hess C, Misurelli S. Studies on bilateral cochlear implants at the University of Wisconsin's Binaural Hearing and Speech Laboratory. J Am Acad Audiol. 2012 Jun;23(6):476-94. doi: 10.3766/jaaa.23.6.9. PMID 22668767
- [Background] Reeder RM, Firszt JB, Holden LK, Strube MJ. A longitudinal study in adults with sequential bilateral cochlear implants: time course for individual ear and bilateral performance. J Speech Lang Hear Res. 2014 Jun 1;57(3):1108-26. doi: 10.1044/2014_JSLHR-H-13-0087. PMID 24686778
- [Background] Spahr AJ, Dorman MF, Litvak LM, Van Wie S, Gifford RH, Loizou PC, Loiselle LM, Oakes T, Cook S. Development and validation of the AzBio sentence lists. Ear Hear. 2012 Jan-Feb;33(1):112-7. doi: 10.1097/AUD.0b013e31822c2549. PMID 21829134

RESULTS

PARTICIPANT FLOW:
Groups:
- Naida Link CROS Device: Individuals 18+ who already have Advanced Bionics CII/90K/Ultra cochlear implants will be given Naida Link Contralateral routing of signal (CROS) device to assess the effect the device has on speech understanding in challenging listening situations and on the quality of life in unilateral cochlear implant recipients and their frequent communication partners.
- Frequent Communication Partners (FCPs): Individuals 18+ who spend at least two hours in-person with Naida Link CROS device users. One FCP will be selected by each CROS device recipient. In this study, A total of seven FCPs were enrolled: six spouses and one mother of the CROS device recipients.
  FCPs will complete a questionnaire to evaluate:
  1. Improvements in communication between themselves and the CROS recipients
  2. Whether these communication improvements affect the FCPs' quality of life.
  No additional data, such as demographics or baseline characteristics, will be collected regarding FCPs as this study focuses on cochlear implant/CROS users.
Period: Overall Study
Arm/Group | Naida Link CROS Device | Frequent Communication Partners (FCPs)
Started | 8 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — This participant didn't meet criteria after screening | 1 | 0

BASELINE CHARACTERISTICS:
Population: 7 Individuals 18+ who already have Advanced Bionics CII/90K/Ultra cochlear implants will be given Naida Link CROS device to assess the effect the device has on speech understanding in challenging listening situations and on the quality of life in unilateral cochlear implant recipients and their frequent communication partners.
Arm/Group | Naida Link CROS Device
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.25 (18.995)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Speech Recognition
Description: AZBio speech testing was performed in a sound booth with two speakers. Sentences at 60 dB were presented in the following conditions: (1) CI-only, speech presented from the front in quiet; (2) CI-only, speech in the non-CI ear in quiet; (3) CI-only, speech in the non-CI ear in noise; (4) CI+CROS device, speech in the non-CI ear in noise. A higher average percentage of words repeated correctly corresponds to greater understanding. The goal was to assess the impact of the CROS device on speech and speech understanding.
  The test was planned at enrollment and after 6 months of CROS use to evaluate long-term effects, but due to COVID-19, only the enrollment test was completed.
Time Frame: At baseline (enrollment visit), with a duration of 50 minutes
Population: 7 participants with unilateral Advanced Bionics CII/90K/Ultra cochlear implant cochlear implant and CROS device
Measure: Mean (Full Range); unit: percentage of words repeated correctly
Groups:
- Cochlear Implant Users: This group comprised of seven Advanced Bionics CII/90K/Ultra cochlear implant recipients who were tested with and without Naida Link contralateral routing of signal (CROS)
  *(within-subjects comparison).
Arm/Group | Cochlear Implant Users
Number analyzed (Participants) | 7
percentage of words repeated correctly
  CI only, with speech presented from front (Quiet environment) | 70.03 [56.83 to 78.52]
  CI only, with speech presented in the non-CI ear (Quiet environment) | 67.92 [50.00 to 90.31]
  CI only, with speech presented in the non-CI ear (Noisy environment) | 30.43 [18.12 to 47.49]
  CI+CROS, with speech presented in the non-CI ear (Noisy environment) | 62.71 [46.08 to 91.74]

2. Secondary Outcome: Auditory Performance and Satisfaction of Cochlear Implant/CROS Device Recipients
Description: The Auditory Performance and Satisfaction Scale for Single-Sided Deafness (APS-SSD) assesses hearing in various environments through 31 statements grouped by context (general, home, social, work/school). Hearing ability is rated from 0: Can function fine to 6: Cannot function at all, lower score indicates better performance.The second section has 2 parts: Part one: 13 statements about satisfaction with CROS device, rated from 0: very satisfied to 6: very dissatisfied, lower score indicates higher satisfaction. Part two: 10 miscellaneous questions regarding overall quality and satisfaction with the CROS device.
  The data table shows the number of subjects reporting improvements in auditory satisfaction, assessed by comparing baseline responses to the 6-month follow-up. A decrease in score indicates perceived improvement. Rows represent categories of participants' auditory experiences, while column shows the number of participants reporting positive changes in that category.
Time Frame: At baseline (enrollment visit) and 6 months after using the CROS device.
Population: Data table is based on the responses of 7 participants with unilateral Advanced Bionics CII/90K/Ultra cochlear implant cochlear implant and CROS device. These participants were assessed for improvements in auditory satisfaction by comparing their responses at baseline and again at the 6-month follow-up. Each row corresponds to a different category/aspect of the participants' auditory experience. The column shows number of participants who reported a positive change for each statement.
Measure: Count of Participants; unit: Participants
Groups:
- Cochlear Implant Users: This group comprised of seven participants who completed the APS-SSD before and after CROS device use (within-subjects comparison).
Arm/Group | Cochlear Implant Users
Number analyzed (Participants) | 7
Participants
  Speech is clearer and easier to understand in a noisy situation | 3
  Speech is clearer and easier to understand in a small group of people | 2
  Speech is clearer and easier to understand when speaking to 1 person in quiet | 5
  Music Sounds better | 6
  Speech sounds more natural | 2
  overall quality of speech is better | 2

3. Secondary Outcome: Frequent Communication Partners' (FCPs) Quality of Life
Description: To asses FCPs' quality of life, they completed the Significant Other Scale for Hearing Disability (SOS-HEAR) questionnaire at baseline and 6 months after the CI users whom they communicate with began using the CROS device. The SOS-HEAR evaluates the disability experienced by the FCP of individuals with hearing loss (i.e., CROS device users). This questionnaire has 26 Statements grouped into: concern for partner, emotional reactions, going out and socializing, relationship changes, communication burden, and communication changes. FCPs rated statements on a 4-point Likert scale ranging from 0-4 with 0=No Problem and 4=A Complete Problem. A lower score represents better outcome.
  Table shows communication outcomes reported by FCPs, assessed by comparing their baseline responses to their 6-month follow-up responses. A decrease in scores represents improvement in communication with CI users. Rows represent communication experience and column shows the count of FCPs within each category
Time Frame: At baseline(enrollment visit), and after 6 months after CROS device use
Population: The table shows communication outcomes reported by 7 Frequent Communication Partners (FCPs) who had at least two hours per week of in-person interactions with the recipient of Advanced Bionics CII/90K/Ultra implants/CROS device
Measure: Count of Participants; unit: Participants
Groups:
- Frequent Communication Partners (FCPs): This group is compromised of 7 Frequent Communication Partners (FCPs) who were enrolled at the same time as the CI users and communicated with them before and after their CROS device use
Arm/Group | Frequent Communication Partners (FCPs)
Number analyzed (Participants) | 7
Participants
  Improved Communication | 5
  No Change in Communication | 1
  Worse Communication | 1

4. Secondary Outcome: Cochlear Implant/CROS Device Recipients' Quality of Life
Description: To evaluate the effect of CROS device use on participant's quality of life, they completed the Nijmegen Cochlear Implant Questionnaire (NCIQ) Adapted from Hinderink et al., 2000, a subjective self-assessment of health-related assessment for cochlear implant (CI) users that includes 60 questions. The answers to the questionnaire range on a 5-point Likert scale never (0), rarely (1), sometimes(3), very often(4), and always (5). A higher score represents a better quality of life experience.
  The table summarizes perceived changes in life quality among participants after 6 months of using the CROS device, assessed by comparing responses at baseline questionnaire to those at the 6-month follow-up. An increase in scores on the questionnaires indicates a perceived improvement in quality of life. Rows represent the categories of life quality changes reported by participants, while the column shows the count of participants within each category.
Time Frame: At baseline, and after 6 months of CROS use
Population: 7 Advanced Bionics CII/90K/Ultra cochlear implant and CROS device users
Measure: Count of Participants; unit: Participants
Groups:
- Naida Link CROS Device: Individuals 18+ who already have Advanced Bionics CII/90K/Ultra unilateral cochlear implants.
  They will be provided with the Naida Link CROS device to evaluate its impact on speech understanding in challenging listening situations. Additionally, they will complete questionnaires and undergo a speech test to assess their speech intelligibility and quality of life.
Arm/Group | Naida Link CROS Device
Number analyzed (Participants) | 7
Participants
  Overall Positive Quality of Life Change | 3
  Overall Negative Quality of Life Change | 2
  Overall No Quality of Life Change | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and other adverse events were not monitored/assessed.
Description: All-cause mortality, serious and other adverse events were not monitored/assessed.
Arm/Group | Naida Link CROS Device
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Questionaries and speech recognition were intended to be measured pre and post-CROS device use. Questionnaires for Cochlear Implant recipients: Modified APS-SSD & Nijmegen, and SOS-HEAR for Frequent Communication Partners were completed after 6 months of CROS device use to assess quality of life. However, due to the COVID-19 pandemic, the speech recognition test was not conducted after 6 months, thereby restricting the evaluation of speech outcomes following prolonged CROS use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT04794179/Prot_SAP_000.pdf